CLINICAL TRIAL: NCT03829553
Title: Hypofractionated Versus Conventional Intensity-Modulated Radiation Therapy for Breast Cancer Patients With an Indication for Regional Nodal Irradiation: A Randomized Multi-center Phase III Trial
Brief Title: Hypofractionated Irradiation At Regional Nodal Area for Breast Cancer Vs Existed Standard Treatment
Acronym: HARVEST
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Collaborators: RenJi Hospital (Other); Shanghai 10th People's Hospital (Other); Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other); Shanghai Zhongshan Hospital (Other); Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other); Affiliated Hospital of Jiangnan University (Other); Cancer Hospital of the University of Chinese Academy of Sciences (Zhejiang Cancer Hospital) (Unknown); The Affiliated Tumor Hospital of Nantong University, Nantong, Jiangsu Province, China (Other)
Responsible Party: Principal Investigator, Jiayi Chen, Chief of Department of Radiation Oncology, Ruijin Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RJBC-HFRNI
Record Dates: First submitted 2019-01-27; First posted 2019-02-04 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2022-05

CONDITIONS: Breast Cancer
Keywords: regional nodal irradiation; IMRT; Hypofractionated radiotherapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Radiation Dose Hypofractionation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypofractionated radiotherapy (Experimental): Patients with an indication for regional nodal irradiation will received 2.67 Gy for 16 fractions to chest wall or whole breast and regional lymph regions (including supraclavicular and internal mammary lymph nodes) and sequential tumor bed boost of 2.67 Gy for 4 fractions following breast conserving surgery
  Interventions: Radiation: Hypofractionated radiotherapy
- Conventional radiotherapy (Active Comparator): Patients with an indication for regional nodal irradiation will received 2 Gy for 25 fractions to chest wall or whole breast and regional lymph regions (including supraclavicular and internal mammary lymph nodes) and sequential tumor bed boost of 2 Gy for 5 fractions following breast conserving surgery.
  Interventions: Radiation: Conventional radiotherapy

INTERVENTIONS:
Radiation: Hypofractionated radiotherapy — 4005 cGy/ 15 fractions / 3 weeks to ipsilateral chest wall or whole breast and regional lymph regions (including supraclavicular and internal mammary lymph nodes) and sequential tumor bed boost of 2.67Gy for 4 fractions in patients with intact breast
  Other Names: Experimental Arm
  Arms: Hypofractionated radiotherapy
Radiation: Conventional radiotherapy — 5000 cGy/ 25 fractions / 5 weeks ipsilateral chest wall or whole breast and regional lymph regions (including supraclavicular and internal mammary lymph nodes) and sequential tumor bed boost of 2Gy for 5 fractions in patients with intact breast
  Other Names: Active Comparator Arm
  Arms: Conventional radiotherapy

SUMMARY:
The main objective of this trial is to investigate the efficacy and safety of hypofractionated radiotherapy of 3 or 4 weeks by comparing with conventional radiotherapy of 5 or 6 weeks using intensity-modulated radiation therapy (IMRT) in breast cancer patients with an indication for regional nodal irradiation (RNI) following mastectomy or breast conserving surgery. Patients will be randomized to hypofractionated radiotherapy or conventional radiotherapy delivered to chest wall or whole breast and regional lymph regions (including supraclavicular and internal mammary lymph nodes). Eligible breast cancer patients will be followed for at least 5 years to evaluate the difference in 5-year locoregional recurrence, over survival, distant metastasis, toxicity and life quality between two groups.

DETAILED DESCRIPTION:
Investigators hypothesize that hypofractionated radiotherapy is equally effective and safe as conventional radiotherapy in breast cancer patients with an indication for regional nodal irradiation. Eligible breast cancer patients are randomized 1:1 into the following two groups: hypofractionated radiotherapy of 2.67 Gy for 16 fractions (and sequential tumor bed boost of 2.67 Gy for 4 fractions in patients with intact breast) and conventional radiotherapy of 2Gy for 25 fractions (and sequential tumor bed boost of 2 Gy for 5 fractions in patients with intact breast). The dose was prescribed to ipsilateral chest wall or whole breast and regional lymph regions (including supraclavicular and internal mammary lymph nodes). All patients are treated with IMRT. The primary endpoint is locoregional recurrence. Patients will be followed at least 5 years after radiotherapy to evaluated over survival, distant metastasis, toxicity and life quality.

ELIGIBILITY:
Inclusion criteria :

* Age 18-75 years old
* unilateral histologically confirmed invasive breast carcinoma of pT1-3
* breast conservation surgery or mastectomy
* Breast reconstruction is allowed
* histologically confirmed positive axillary lymph nodes (positive sentinel lymph nodes without axillary dissection is allowed)
* Life expectancy of >5 years
* A minimum negative surgical margin width of >2mm
* Karnofsky Performance Status ≥80
* Estrogen-receptor, Progesterone-receptor, human epidermal growth factor receptor-2 (HER-2) and Ki67 index can be performed on the primary breast tumor or axillary nodes.
* Written informed consent

Exclusion criteria:

* Supraclavicular lymph nodes, positive ipsilateral internal mammary lymph nodes or residual axillary nodes that may be eligible for a boost dose.
* Pregnant or lactating
* Severe non-neoplastic medical comorbidities
* Diagnosis of non-breast malignancy within 5 years preceding enrollment (except for basal cell carcinoma of the skin or carcinoma in situ of the cervix).
* Simultaneous contralateral breast cancer
* Previous RT to thoracic and/or axillary, cervical region
* Active collagen vascular disease
* Evidence of distant metastatic disease and/or T4 disease

Notes for exlusion criteria:

1. Patients with severe non-neoplastic medical comorbidities (e.g.,severe ischemic heart disease, severe arrhythmia or severe chronic obstructive pulmonary disease ) that would preclude radiation treatment will be excluded.
2. Simultaneous contralateral breast cancer includes histologically confirmed DCIS only.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 801 (Estimated)
Dates: Start 2019-02-21 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Locoregional recurrence (LRR) | 5 years
  any first recurrence confirmed by histology or cytology in the ipsilateral chest wall or breast or regional nodes areas (including axillary, supraclavicular, infraclavicular lymph nodes or IMN)

SECONDARY OUTCOMES:
Distant metastasis free survival (DMFS) | 5 years
  the time from the date of randomization to any recurrence of tumor at distant sites or death from any cause.
Invasive recurrence-free survival (IRFS) | 5 year
  the time from the date of randomization to any invasive recurrence of tumor, distant metastases or death from any cause and second invasive primaries, including invasive neoplasms of the breast.
over survival (OS) | 5 years
  the time from the date of randomization to the date of death from any cause or end of the follow-up.
Number of Participants with excellent or good Cosmetic outcomes following breast conserving surgery-Harvard/NSABP/RTOG scoring scale | 5 years
  The time from the date of randomization to 5 years after completion of radiotherapy, the cosmetic outcomes will be evaluated before radiotherapy, every week during radiotherapy, 4 weeks after the last fraction received, every 6 months during the first 2 years and annually thereafter. The cosmetic outcomes are evaluated based on the Allegheny General Modification of the Harvard/(National Surgical Adjuvant Breast and Bowel Project) NSABP/ (Radiation Therapy Oncology Group) RTOG scoring scale which graded patients into the following four classifications: excellent, when compared to the untreated breast, there is a minimal or no difference in the size or shape of the treated breast; good, slight difference in the size or shape of the treated breast; fair, obvious difference in the size or shape of the treated breast; and poor, marked change in the size or shape of the treated breast.
Number of Participants with ≥Grade1 Acute Radiation-induced Toxicity | 6 months
  within time from beginning of RT to 6 months after completion of RT assessed according to the Common Terminology Criteria for Adverse Events (CTCAE) version 3.0.
Number of Participants with ≥Grade1 Late Radiation-induced Toxicity | 5 years
  within time from 6 months after completion of RT to 5 years after completion of RT assessed according to the RTOG/ European Organization for Research on Treatment of Cancer (EORTC） Late Radiation Morbidity Scoring Schema and CTCAE version 3.0
Reconstruction complications | 5 years
  number of participants with any reconstruction complications (flap necrosis, capsular contracture, infection, loss of implant/expander or flaps, et al) and the interval between the RT and reconstruction complications will be recorded. Patient reported outcome with reconstruction will be evaluated by Breast-Q questionnaires before RT and 12 months after RT.

OTHER OUTCOMES:
Quality of Life-EORTC QLQ-C30 | 1 years
  The time from the date of randomization to 5 years after completion of radiotherapy, Quality of life will be assessed before radiotherapy, every week during radiotherapy, 4 weeks after the last fraction received, every 6 months during the first 2 years and annually thereafter using self-administered questionnaire EORTC QLQ-C30
Quality of Life-EORTC QLQ-C30 | 5 years
  The time from the date of randomization to 5 years after completion of radiotherapy, Quality of life will be assessed before radiotherapy, every week during radiotherapy, 4 weeks after the last fraction received, every 6 months during the first 2 years and annually thereafter using self-administered questionnaire EORTC QLQ-C30
Quality of Life-EORTC QLQ-BR23 | 1 years
  The time from the date of randomization to 5 years after completion of radiotherapy, Quality of life will be assessed before radiotherapy, every week during radiotherapy, 4 weeks after the last fraction received, every 6 months during the first 2 years and annually thereafter using self-administered questionnaire EORTC QLQ-BR23
Quality of Life-EORTC QLQ-BR23 | 5 years
  The time from the date of randomization to 5 years after completion of radiotherapy, Quality of life will be assessed before radiotherapy, every week during radiotherapy, 4 weeks after the last fraction received, every 6 months during the first 2 years and annually thereafter using self-administered questionnaire EORTC QLQ-BR23

CONTACTS AND LOCATIONS:
Overall Officials: Jia-Yi Chen, Study Chair — Ruijin Hospital
Locations (1):
- Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Xie J, Xu F, Zhao Y, Cai G, Lin X, Zhu Q, Lin Q, Yao Y, Xu C, Cai R, Wang S, Tang X, Chen C, Zheng S, Chen M, Chen M, Qian X, Shen C, Li J, Xu H, Xu F, Han Y, Li M, Ou D, Shen KW, Qi WX, Cao L, Huang X, Chen J. Hypofractionated versus conventional intensity-modulated radiation irradiation (HARVEST-adjuvant): study protocol for a randomised non-inferior multicentre phase III trial. BMJ Open. 2022 Sep 1;12(9):e062034. doi: 10.1136/bmjopen-2022-062034. PMID 36581983